CLINICAL TRIAL: NCT00641381
Title: High Dose Chemotherapy and Combination Anti-HIV Therapy for HIV-Associated Hodgkin's and Non-Hodgkin's Lymphoma
Brief Title: Carmustine, Etoposide, Cyclophosphamide, and Stem Cell Transplant in Treating Patients With HIV-Associated Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99067; P30CA033572 (NIH); CHNMC-99067; CDR0000589621 (Registry Identifier: NCI PDQ); NCI-2010-00431 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-03-21; First posted 2008-03-24 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Lymphoma
Keywords: stage III adult Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent mantle cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; AIDS-related diffuse large cell lymphoma; AIDS-related diffuse mixed cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related lymphoblastic lymphoma; AIDS-related small noncleaved cell lymphoma; Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; HIV Infections; Treatment Experienced
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Mantle-Cell; Recurrence; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; HIV Infections | interventions — Carmustine; Cyclophosphamide; Etoposide; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (high-dose chemotherapy, anti-HIV therapy) (Experimental): Patients undergo leukapheresis to obtain PBSCs for transplantation. At least 5 days later, patients with an adequate number of collected cells proceed to high-dose chemotherapy. Patients receive carmustine IV over 4 hours on days -7 to -5, etoposide IV over 4 hours on day -4, and cyclophosphamide IV on day -2. Patients receive an autologous PBSC infusion on day 0.
  Interventions: Drug: carmustine; Drug: cyclophosphamide; Drug: etoposide; Other: pharmacological study; Procedure: autologous hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Drug: carmustine — 150 mg/m2 day -7, -6,and -5 prior to stem cell reinfusion
Drug: cyclophosphamide — 100 mg/kg on day -2 prior to stem cell reinfusion
Drug: etoposide — 60 mg/kg on day -4 prior to stem cell reinfusion
Other: pharmacological study — Prior to start of etoposide infusion, 2 hours after start of infusion, just prior to the end of infusion, then at 0.5, 1, 2, 4, 24 and 48 hours after the end of infusion
Procedure: autologous hematopoietic stem cell transplantation — Reinfusion of autologous stem cells
Procedure: peripheral blood stem cell transplantation — Reinfusion of autologous stem cells

SUMMARY:
RATIONALE: Giving high-dose chemotherapy drugs, such as carmustine, etoposide, and cyclophosphamide, before a peripheral blood stem cell transplant stops the growth of cancer cells by stopping them from dividing or killing them. After treatment, stem cells that were collected from the patient's blood are returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy.

PURPOSE: This clinical trial is studying the side effects of giving high-dose carmustine, etoposide, and cyclophosphamide together with a stem cell transplant and to see how well it works in treating patients with HIV-associated lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the feasibility and toxicity of high-dose chemotherapy comprising carmustine, etoposide, and cyclophosphamide followed by autologous stem cell infusion in patients with HIV-associated lymphoma receiving combination anti-HIV therapy and to determine the efficiency of stem cell collection from these patients.
* To estimate the disease-free and overall survival of patients treated with this regimen.
* To evaluate HIV viral load, CD+4/CD+8 counts, and immune recovery after high-dose anti- lymphoma chemotherapy.
* To determine the pharmacokinetics of high-dose etoposide in patients receiving highly active anti-retroviral therapy (HAART).

OUTLINE: Patients undergo leukapheresis to obtain peripheral blood stem cells (PBSCs) for transplantation. At least 5 days later, patients with an adequate number of collected cells proceed to high-dose chemotherapy.

* High-dose chemotherapy: Patients receive carmustine IV over 4 hours on days -7 to -5, etoposide IV over 4 hours on day -4, and cyclophosphamide IV on day -2.
* Autologous PBSC transplantation: Patients receive PBSC infusion on day 0. Patients undergo blood sample collection periodically for pharmacokinetic studies of etoposide.

After completion of study treatment, patients are followed at approximately 30 days and 100 days, every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* HIV seropositive at or before the time of lymphoma diagnosis
* Subjects must be on a multi-drug regimen (excluding azidothymidine) to maintain HIV viral load less than 50,000 Gc/mL; if the CD4 count at enrollment is less than 100 then the viral load should be less than 10,000 by reverse transcriptase polymerase chain reaction (Rt-PCR); if the CD4 count is greater than 100/mm^3 prior to the start of any lymphoma chemotherapy and is greater than 100/mm^3 for at least 3 months then the viral load must be less than 150,000 gc/ml and clinically stable; if no pre-chemotherapy CD4 counts are available, then viral load alone will be used from enrollment
* The known hematopoietic toxicity of AZT (zidovudine) prohibits its use pre-transplant during stem cell collection and during the immediate period of engraftment post-transplant; resumptions of AZT should not begin until there is evidence of stable engraftment; therefore, AZT should not be resumed until at least 2 months after last blood product support is used; since platelet support continues until approximately day +14 days in our experience with acquired immune deficiency syndrome (AIDS) patients transplanted date, AZT will be prohibited until at least 2 months after transplant; therefore, if the anti-HIV drug combination needs to be modified then AZT can be part of the new regimen
* Karnofsky performance status >= 70%
* Biopsy proven intermediate grade or high-grade Non-Hodgkin's lymphoma, (working formulation groups D-H and J, and Plasmablastic lymphoma of any disease state, including first remission given the poor risk nature of this histology) or Hodgkin's lymphoma of any subtype except nodular lymphocytic and histiocytic (L&H) lymphocyte predominant; tissue histology will be reviewed at the City of Hope
* Patients with prior marrow involvement must demonstrate < 10% involvement (by morphology) pre stem cell collection
* Pretreatment serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvate transaminase (SGPT) < 1.5 x institutional upper limit of normal
* Serum bilirubin < 1.5 x institutional upper limit of normal
* Patients who are Hepatitis C antibody positive or Hepatitis B surface antigen positive without clinical evidence of cirrhosis will be eligible after further evaluation; specifically, if patient hepatitis C or B positive viral loads will be measured; patients with hepatitis B and ongoing evidence of viral replication may require therapy prior to receiving high dose chemotherapy; this decision will be at the discretion of the treating physician
* Serum creatinine < 2 x institutional upper limit of normal and a 24 hour urine creatinine clearance > 60 cc/min
* Prothrombin time (PT)/partial thromboplastin time (PTT) < 2 x normal
* Forced expiratory volume in one second (FEV1) or diffusing capacity of the lung for carbon monoxide (DLCO) >= 50% predicted
* Left ventricular ejection fraction (LVEF) >= 50% (by 2 dimensional [2 D] echocardiogram or multi gated acquisition scan [MUGA] scan); absence of cardiomyopathy, congestive heart failure or dysrhythmia
* If female of child bearing potential, must have negative serum pregnancy test
* Subjects must be on a prophylactic regimen for pneumocystis pneumonia if the CD4 counts are < 200
* Subjects who are not in complete remission must have measurable disease; measurable disease means that there are bidimensionally measurable lesions with clearly defined margins using either a medical photograph, computerized axial tomography (CAT) scan or magnetic resonance imaging (MRI) scan, or palpation of lesions with both diameters >= 2 cm; evaluable disease means that the lesions are only unidimensionally measurable, or have indistinct margins or have both diameters < 0.5 cm, or that the palpable lesions have a diameter < 2.0 cm, or are lesions in bone; pleural effusions and ascites are considered nonevaluable disease; scans must be within 28 days from enrollment
* A minimum of 2.5 x 10^6 CD34 cells/kg must have been collected
* Hodgkin's Lymphoma:

  * Partial response after standard chemotherapy OR
  * First relapse after initial complete remission with standard chemotherapy
* Non-Hodgkin's Lymphoma:

  * First complete remission after standard chemotherapy with high risk features as specified by the International Prognostic Index;
  * Partial response after standard chemotherapy; OR
  * Relapse after initial complete remission with standard chemotherapy

Exclusion Criteria:

* Active bacterial or fungal infection
* AIDS related opportunistic infection within past year, excluding treatment-responsive Mycobacterium Avium Intracellular infection, and treatment-responsive oral thrush, herpes simplex or herpes zoster
* Active cytomegalovirus (CMV) retinitis or other CMV-related organ dysfunction; patients with a history of treated CMV infection are not excluded
* Relapse of pneumocystis carinii pneumonia within the past year
* AIDS related syndromes or symptoms that pose a perceived excessive risk for transplantation-related morbidity as determined by the principle investigator
* Intractable and severe diarrhea as defined as > 1500 cc diarrheal fluid per day of diarrhea causing persistent severed electrolyte abnormalities or hypoalbuminemia
* History of grade III hemorrhagic cystitis due to prior chemotherapy
* Pregnant or nursing women
* Any prior malignancy except treated basal cell carcinoma of the skin; females with cervical dysplasia may be included at the discretion of the treating physician and the principle investigator
* Patients with a history of positive cerebrospinal fluid (CSF) cytology that has become negative with intrathecal chemotherapy are eligible; patients should have a negative spinal fluid cytology within thirty days prior to enrollment
* Abnormal cytogenetics on screening bone marrow biopsy
* Psychosocial conditions that hinder compliance

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2000-05-10 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Number of days to engraftment as defined by the standard operating procedures of the department of biostatistics at the City of Hope | Day 100 post stem cell reinfusion
Feasibility and treatment-associated toxicity of this regimen | 1 year post stem cell reinfusion

SECONDARY OUTCOMES:
Ability to mobilize adequate numbers of peripheral blood stem cells (2.5 x 10e6 CD34+cells) | At the completion of stem cell collection
Disease-free and overall survival | 2 years post stem cell reinfusion
HIV viral load, CD4+/CD8+ counts, and immune recovery | 2 years post stem cell reinfusion

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Y. Krishnan, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States